CLINICAL TRIAL: NCT07025057
Title: Multilevel Community-centered Intervention to Reduce Pregnancy Related and Associated Morbidity and Mortality (PRAMM) Disparities in Non-Hispanic Black and Hispanic Medicaid-insured Individuals
Brief Title: Multilevel Community-Centered Intervention to Reduce Pregnancy Related and Associated Morbidity and Mortality (PRAMM) Disparities
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Michigan State University (Other)
Collaborators: Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH)
Responsible Party: Principal Investigator, Cristian Meghea, Associate Professor, Michigan State University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Health Services Research
Other Study IDs: STUDY00009358; U54HD113291 (NIH)
Record Dates: First submitted 2025-06-02; First posted 2025-06-17 (Actual); Last update posted 2025-06-17 (Actual); Status verified 2025-06

CONDITIONS: Provider Confidence; Provider Behavior
Keywords: Maternal mortality; Maternal morbidity
MeSH Terms: conditions — Maternal Death

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Provider training (Experimental): The providers in this arm will receive training
  Interventions: Behavioral: Provider training

INTERVENTIONS:
Behavioral: Provider training — The study will address patient-provider interactions through actionable, experiential provider trainings focused on communication provider, cultural relevance, and awareness of and referrals to community care services including Community Health Workers (CHW) and home visiting, for both clinical and community settings. Trainings are rooted in both history and in current research about how to address maternal mortality disparities, and will include self-learning, didactics, reflection, discussion, and identifying ways to tailor trainees settings to better hear, respect, and meet the needs of perinatal Black and Hispanic women.

SUMMARY:
The goal of the study involving human subjects is to train providers to address patient-provider interactions. The study will survey providers to assess pre-post knowledge, understanding, and behavior changes.

DETAILED DESCRIPTION:
Provider/practice level intervention. The study will address patient-provider interactions through actionable, experiential provider trainings focused on communication provider, cultural relevance, and awareness of and referrals to community care services including CHWs and HV, for both clinical and community settings. Trainings are rooted in both history and in current research about how to address maternal mortality disparities, and will include self-learning, didactics, reflection, discussion, and identifying ways to tailor trainees settings to better hear, respect, and meet the needs of perinatal NHB/H women.

ELIGIBILITY:
Inclusion Criteria:

* Providing care to pregnant and postpartum women in Wayne, Kent, and Genesee Counties in MI

Exclusion Criteria:

* None

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 480 (Estimated)
Dates: Start 2025-02-03 (Actual); Primary Completion 2029-08-01 (Estimated); Study Completion 2030-08-15 (Estimated)

PRIMARY OUTCOMES:
Provider confidence. Assessed through questionnaire. | Assessment immediately after the provider training intervention
  Pre-post intervention change in provider confidence regarding provider-patient interactions

CONTACTS AND LOCATIONS:
Overall Officials: Cristian Meghea, PhD, Principal Investigator — Michigan State University
Locations (1):
- Strong Beginings, Grand Rapids, Michigan, United States

IPD SHARING:
Plan to Share IPD: Yes
The study is collecting data and later will be sharing project-generated data according to NIH's requirements for depositing relevant de-identified data into appropriate NIH data archives.